## **CONSENT FORM**

Physiological and sensory responses to prolonged fasting in humans
Mr Harry Smith (H.A.Smith@bath.ac.uk); Professor James Betts (J.Betts@bath.ac.uk)

## Please initial box if you agree with the statement

| 1. | have been provided with information explaining what participation in this project involves | |
|---|---|---|
| 2. | I have had an opportunity to ask questions and discuss this project. | |
| 3. | I have received satisfactory answers to all questions I have asked. | |
| 4. | I have received enough information about the project to make a decision about my participation. | |
| 5. | I understand that I am free to withdraw my consent to participate in the project up until the final measure of the final trial without having to give a reason for withdrawing. | |
| 6. | I understand that I am free to withdraw my data within two week | s of my participation. |
| 7. | I understand the nature and purpose of the procedures involved in this project (e.g. fasting for ~82 hours, providing muscle and fat samples before and after the fast, meal testing). These have been communicated to me on the information sheet accompanying this form. | |
| 8. | I understand and consent to my RNA (genetic information) being analysed and used in this study. | |
| 9. | I understand and acknowledge that the investigation is designed to promote scientific knowledge and that the University of Bath will use the data I provide only for the purpose(s) set out in the information sheet. | |
| 10 | I understand the data I provide will be treated as confidential, and that on completion of the project my name or other identifying information will not be disclosed in any presentation or publication of the research. | |
| 11. I understand that my consent to use the data I provide is conditional upon the University complying with its duties and obligations under the Data Protection Act. | | |
| 12 | . I hereby fully and freely consent to my participation in this project | ct. |
| | Participant's signature: Participant name in BLOCK Letters: Researcher's signature: Researcher name in BLOCK Letters: | <br>_Date: |

If you have any concerns or complaints related to your participation in this project please direct them to the Secretary of the Research Ethics Approval Committee for Health, Rebecca Wise (r.wise@bath.ac.uk, 01225 384714)